CLINICAL TRIAL: NCT05859477
Title: Nivolumab and CAPOX in Patients With FGFR2/PD-L1-positive Metastatic Gastric Adenocarcinoma: a Single-arm, Phase 2 Study
Brief Title: Nivolumab in Combination With Chemotherapy for FGFR2-positive Metastatic Gastric Cancer
Acronym: NIVOFGFR2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kidney Cancer Research Bureau (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIVOFGFR2
Record Dates: First submitted 2023-05-01; First posted 2023-05-16 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Metastatic Gastric Cancer; PD-L1 Gene Amplification; FGFR2 Amplification
MeSH Terms: conditions — Stomach Neoplasms | interventions — Nivolumab; Capecitabine; Oxaliplatin

STUDY DESIGN:
Intervention Model Description: Nivolumab in combination with chemotherapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nivolumab in combination with chemotherapy (Experimental): Nivolumab 360 mg with CAPOX (capecitabine and oxaliplatin) every 3 weeks
  Interventions: Drug: Nivolumab; Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Nivolumab — 360 mg, i.v., every 3 weeks
  Other Names: Opdivo
Drug: Capecitabine — capecitabine 1000 mg/m², orally, twice a day, days 1-14 of each cycle
  Other Names: Xeloda
Drug: Oxaliplatin — 130 mg/m², i.v., day 1, every 3 weeks

SUMMARY:
The goal of this phase 2 clinical trial is to evaluate the efficacy of nivolumab in combination with CAPOX in patients with FGFR2-positive/PD-L1-positive/HER2-negative metastatic gastric cancer.

DETAILED DESCRIPTION:
On April 16, 2021, the Food and Drug Administration approved first-line therapy with nivolumab and fluoropyrimidine-platinum-containing chemotherapy for metastatic gastric adenocarcinoma. Patients with PD-L1 expression benefit the most from this treatment.

Fibroblast growth factor receptor 2 (FGFR2) is a predictor of poor overall survival and a potential target for targeted therapy. However, there is no data of nivolumab efficacy in patients with combined expression of PD-L1 and FGFR2.

The aim of this study is to evaluate the preliminary efficacy of nivolumab in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated, unresectable advanced or metastatic gastric adenocarcinoma
* Measurable lesions according to the RECIST 1.1 criteria
* PD-L1 Combined Positive Score (CPS) of five or more assessed by Dako PD-L1 immunohistochemistry 28-8 pharmDx assay
* Positive FGFR2 overexpression status by immunohistochemistry defined as exhibiting any moderate (2+) to strong (3+) membranous staining in more than 1% of tumor cells
* Possibility to assess the amplification of FGFR2
* HER2-negative status
* ECOG PS 0-2
* Age >= 18 years old
* Adequate function of organs
* Absence of any psychological, family, social or geographical circumstances that could potentially serve as obstacles to the implementation of the study
* Signed Informed Consent

Exclusion Criteria:

* Participation in another clinical study and concomitant treatment with any research drug or any study of antitumor therapy, including radiation, within 28 days before inclusion in this study
* Presence of metastases in the central nervous system and / or carcinoma of the meninges at the time of inclusion in the study
* Presence or history of present signs of any condition, therapy or laboratory abnormalities that could limit the interpretation of the results of this study
* Any malignant tumor within the previous 5 years, with the exception of adequately cured cervical cancer in situ or squamous cell skin cancer, or basal cell skin cancer with limited growth, subject to adequate control over the course of this disease
* Pregnancy
* Known positive status for human immunodeficiency virus (HIV) or active hapatitis B and C
* Surgery within 7 days before the first dose of the study drug
* Signs of bleeding or hemorrhagic diathesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2022-06-05 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
1-year progression-free survival (PFS) | 12 months
  Proportion of patients who will be progression-free at 1 year

SECONDARY OUTCOMES:
Median PFS | 18 months
  From first day of treatment to the first observation of disease progression or death due to any cause
Median overall survival (OS) | 24 months
  From first day of treatment to time of death due to any cause.
Objective response rate (ORR) | 18 months
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Toxicity Summary | Up to 30 days post treatment
  toxicity assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Grade 3 and above adverse events possibly, probably or definitely related to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ilya Tsimafeyeu, Study Chair — Bureau for Cancer Research
Locations (1):
- Bureau for Cancer Research, New York, New York, United States